CLINICAL TRIAL: NCT00925847
Title: Open Multicenter Study of Lithium in Patients With Amyotrophic Lateral Sclerosis LISLA
Brief Title: Effect of Lithium Carbonate in Patients With Amyotrophic Lateral Sclerosis
Acronym: LISLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P080401
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2009-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Lithium; Survival
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: lithium

INTERVENTIONS:
Drug: lithium — lithium LP 400mg daily po (doses were adjusted during the study to maintain targeted blood levels.)

SUMMARY:
The purpose of the study is to determine whether lithium is safe and effective in the treatment of ALS

DETAILED DESCRIPTION:
Daily doses of lithium, have been found to delay progression of amyotrophic lateral sclerosis (ALS) in a 15-month study of 44 patients with ALS. At the end of the trial, about 30 percent of the patients that took riluzole had died, while all those receiving riluzole plus lithium had survived. the lithium group had slower progression as measure by a test of breathing (FVC) and strength.

This study will determine whether lithium in combination with riluzole delay progression of patients with amyotrophic lateral sclerosis disease in comparison of an historical cohort of ALS patients treated with riluzole alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically possible, clinically probable laboratory-supported, clinically probable or clinically definite ALS (according to WNF EL Escorial diagnostic criteria, revised according to the AIRLIE House Conference 1998)
* Concomitant standard Riluzole therapy (50mg twice daily)
* patients included in ALS reference center
* women of childbearing age be non-lactating and surgically sterile or using a highly effective method of birth control and have a negative pregnancy test
* capable of thoroughly understanding all information given and giving full informed consent according to GCP
* Patients with gastrostomy

Exclusion Criteria:

* evidence of major psychiatric disorder or clinically evident dementia precluding evaluation of symptoms
* any medical condition known to contre-indicate lithium treatment (dysthyroid, cardiopathy, renal insufficiency)
* presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment
* known hypersensitivity to any component of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Survival in patients with ALS treated with lithium and riluzole compared to historical cohort (patients treated with riluzole alone ) | 15 months

SECONDARY OUTCOMES:
Functional Assessment Change in ALS Functional Rating Score (ALSFRS-R slope) | 15 months
Muscle Strength Change in MMT score (MMT slope) | 15 months
Rate of decline of respiratory function determined as SVC over the 15 month treatment period | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Lucette Lacomblez, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France